CLINICAL TRIAL: NCT04012541
Title: A Randomized Control Trial of Comprehensive Oral Intervention in Patients With Acute Myocardial Infarction: a Pilot Study
Brief Title: Comprehensive Oral Intervention in Patients With AMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, Si-Hyuck Kang, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AMI oral intervention
Record Dates: First submitted 2019-06-14; First posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Acute Myocardial Infarction; Dental Diseases
MeSH Terms: conditions — Stomatognathic Diseases

STUDY DESIGN:
Intervention Model Description: This study is randomized controlled trial. Patients who agreed to the study were randomly assigned to the intervention group and control group at a 1: 1 ratio.
Who Masked: Investigator
Masking Description: Participating patients and dentists are not able to blind information about random allocation. However, in order to reduce the bias, the cardiologist who treats the patient and prescribes the medicines performs an investigator-masked design that masks information about the treatment group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): 1. post-myocardial infarction management
  2. basic periodontal examinations
  3. active dental procedure
  Interventions: Procedure: active dental procedure; Drug: post-myocardial infarction management; Radiation: basic periodontal examinations
- control group (Active Comparator): 1. post-myocardial infarction management
  2. basic periodontal examinations
  Interventions: Drug: post-myocardial infarction management; Radiation: basic periodontal examinations

INTERVENTIONS:
Procedure: active dental procedure — scaling and root planing
  Arms: treatment group
Drug: post-myocardial infarction management — aspirin, clopidogrel, ticagrelor
  Other Names: dual antiplatelet drug
Radiation: basic periodontal examinations — panorama radiograph : full mouth periapical radiograph

SUMMARY:
The investigators performed a randomized controlled trial with investigator-masked design enrolling subjects with acute myocardial infarction.

The purpose of this study is to find a treatment strategy to reduce the risk of recurrence of myocardial infarction through oral hygiene improvement.

DETAILED DESCRIPTION:
Subjects were divided into a treatment group and a control group. Both sides receive basic periodontal examinations, but the treatment group receives active dental procedure such as scaling and root planing. Both groups also receive post-myocardial infarction management.

As part of a pilot study, this study used the primary outcome measure for changes in surrogate markers rather than clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18
* Patients diagnosed with type 1 or 2 MI according to the Fourth Universal Definition of Myocardial Infarction (2018) criteria
* Patients with baseline hsCRP (high-sensitivity C-reactive protein) elevated above 1.0 mg / dL

Exclusion Criteria:

1. clinical exclusion criteria

   * Inability to provide informed consent
   * Patients who are predicted to have low compliance
   * Those whose life expectancy is less than 3 months due to cardiovascular disease or other reasons
   * Those who are considered to be too poor condition to perform dental treatment or have a high risk of bleeding
   * Those who need active dental treatment such as extraction
   * Patients suspected of having active infection
   * Those who are taking long-term systemic antibiotics or receiving immunosuppressive treatment
2. periodontal exclusion criteria

   * Fully edentulous (Except for fixed implant restorations)
   * If more than 15 teeth and implants do not exist
   * If the last dental visit experience is less than 6 months
   * If periodontal treatment is not possible by the researcher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2019-07-05 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
hsCRP | at 3 months
  hsCRP(high sensitivity C-reactive protein), mg/dL

SECONDARY OUTCOMES:
surrogate blood markers | at 3 months
  FBS & Total cholesterol & LDL-cholesterol & HDL-cholesterol & Triglyceride & Apolipoprotein A & Apolipoprotein B, mg/dL
patient symptom | at 3 months & 12 months
  NYHA functional class
Systolic & diastolic blood pressure | at 3 months & 12 months
  automated blood pressure, mmHg
Exercise performance | at 3 months
  Treadmill test
Death | at 12 months
  number of cardiovascular death
unscheduled coronary revascularization | at 12 months
  number of unscheduled coronary revascularization
stroke | at 12 months
  number of stroke
HF admission | at 12 months
  number of HF admission
unstable angina | at 12 months
  number of unstable angina
recurrent MI | at 12 months
  number of recent MI

CONTACTS AND LOCATIONS:
Overall Officials: Si-Hyuck Kang, MD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ye Z, Cao Y, Miao C, Liu W, Dong L, Lv Z, Iheozor-Ejiofor Z, Li C. Periodontal therapy for primary or secondary prevention of cardiovascular disease in people with periodontitis. Cochrane Database Syst Rev. 2022 Oct 4;10(10):CD009197. doi: 10.1002/14651858.CD009197.pub5. PMID 36194420